CLINICAL TRIAL: NCT03092817
Title: A Randomized Double Blind Placebo Controlled Trial of Adjunctive Dexamethasone for the Treatment of HIV-infected Adults With Tuberculous Meningitis
Brief Title: Adjunctive Corticosteroids for Tuberculous Meningitis in HIV-infected Adults (The ACT HIV Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Pham Ngoc Thach Hospital, Ho Chi Minh City, Vietnam (Other); Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other); Dr Cipto Mangunkusumo General Hospital (Other); RSUP Persahabatan Hospital, Jakarta, Indonesia (Unknown); Oxford University Clinical Research Unit Indonesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 26TB
Record Dates: First submitted 2017-03-15; First posted 2017-03-28 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Tuberculosis; Tuberculous Meningitis; Drug-Induced Liver Injury; HIV; IRIS
Keywords: Tuberculosis; tuberculous meningitis; drug induced liver injury; HIV; IRIS; randomized controlled trial; dexamethasone
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Meningeal; Chemical and Drug Induced Liver Injury | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Active Comparator): standard anti-tuberculosis drugs plus dexamethasone for 6-8 weeks
  Interventions: Drug: Dexamethasone
- Identical placebo (Placebo Comparator): standard anti-tuberculosis drugs plus placebo for 6-8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Active treatment with dexamethasone from randomisation (IV followed by oral according to disease severity at the start of treatment): dexamethasone for intravenous injection and dexamethasone for oral ingestion
  Arms: Dexamethasone
Other: Placebo — Treatment with matched placebo:
  Standard saline for intravenous injection and placebo oral tablets containing cellulose
  Arms: Identical placebo

SUMMARY:
The investigators will conduct a randomized, double blind, placebo controlled trial of adjunctive dexamethasone in the initial (6-8 weeks) treatment of tuberculous meningitis in Vietnamese adults. The trial will address a primary hypothesis in all enrolled patients, and a secondary hypothesis in a sub-group of enrolled patients who develop anti-tuberculosis drug-induced liver injury (DILI). The primary hypothesis is adjunctive dexamethasone increases survival from TBM in HIV co-infected adults. The secondary hypothesis is current guidelines for the management of anti-tuberculosis drug-induced liver injury in those with TBM result in the premature interruption of rifampicin and isoniazid (the critical active drugs in early therapy) and are thereby placing participants at risk of poor outcomes.

DETAILED DESCRIPTION:
Mycobacterium tuberculosis causes ~9 million new cases of tuberculosis and ~1.5 million deaths annually, around 0.4 million of whom are co-infected with HIV. Tuberculous meningitis (TBM) is the most severe form of tuberculosis, killing around 30% of all sufferers despite appropriate anti-tuberculosis chemotherapy. It is especially common in young children, and in those infected with HIV.

There is a longstanding hypothesis that death from TBM results from an excessive intracerebral inflammatory response. The corollary of this hypothesis has been that adjunctive anti-inflammatory treatment with corticosteroids (e.g. dexamethasone) improves survival, which has been demonstrated in predominantly HIV-uninfected individuals in a small number of trials. Yet how corticosteroids improve survival, and whether they do so in HIV-infected patients, remains uncertain. The primary objective of this trial is to determine whether or not adjunctive corticosteroids reduce deaths from TBM in HIV-infected adults.

Adjunctive dexamethasone might improve outcomes from HIV-associated TBM by diverse mechanisms. First, it may control the early intracerebral inflammatory response, reducing cerebral oedema and intra-cranial pressure. Second, it may prevent the potentially life-threatening complications of hydrocephalus, infarction and tuberculoma formation. Third, it may prevent the incidence of anti-retroviral (ARV) treatment-associated neurological immune reconstitution inflammatory syndrome (IRIS). Finally, dexamethasone may help reduce the risk of drug-induced liver injury and thereby improve outcome by enabling uninterrupted anti-tuberculosis treatment.

The current evidence-base for using adjunctive corticosteroids for the treatment of HIV-associated TBM is restricted to 98 adults recruited to a trial in Vietnam published in 2004. This trial randomized a total of 545 subjects (98 of them HIV-positive) and reported an overall reduction in 9-month mortality due to dexamethasone from 41.3% (112/271) to 31.8% (87/274) (hazard ratio of time to death 0.69; 95% CI 0.52-0.92, P=0.01). While there was no clear evidence of treatment effect heterogeneity according to HIV status, the number of included HIV-infected subjects was low and the observed benefit in that subgroup was smaller: 61.4% (27/44) in the dexamethasone group died, compared to 68.5% (37/54) in the placebo group (hazard ratio of time to death 0.86; 95% CI 0.52-1.41; P=0.55).

There are limited data from HIV-infected patients with TBM treated with dexamethasone, but findings from studies using corticosteroids in HIV-infected individuals with other forms of tuberculosis and other opportunistic infections suggest corticosteroids may cause harm in those with advanced HIV infection. There is evidence that corticosteroids may increase the risk of HIV-associated malignancies, especially Kaposi sarcoma. Furthermore, a recent trial of adjunctive dexamethasone for HIV-associated cryptococcal meningitis performed in Southeast Asia and Africa found dexamethasone was associated with worse outcomes, with increased risk of secondary infections, hyperglycaemia and electrolyte abnormalities, and disability.

On the basis of these limited data most international guidelines cautiously recommend dexamethasone should be given for HIV-associated TBM, but all acknowledge the paucity of evidence and the need for additional controlled trial data. Our trial will meet the need for more data and aims to provide definitive evidence as to the risk/benefit of adjunctive dexamethasone in the treatment of this important and very severe disease.

Our secondary objective is to investigate alternative management strategies in a subset of patients who develop drug-induced liver injury that will enable the safe continuation of rifampicin and isoniazid therapy whenever possible. The investigators will perform an open, randomised comparison of three management strategies with the aim of demonstrating which strategy results in the least interruption in R and H treatment. All patients enrolled in the trial will be eligible to take part in this study, with the exception of those known to have TBM caused by isoniazid resistant or MDR M. tuberculosis. Consent will be sought at enrolment, with an option given to patients to enrol in the main study, but not the 'drug-induced liver injury strategy study'.

Eligible patients will be randomised to one of three strategies:

1. Observe: measure transaminases, bilirubin, and INR every 3 days; do not change/stop anti-tuberculosis drugs unless transaminases rise to ≥10x normal, or total bilirubin rises >2.0mg/dl (>34 µmol/L), or INR >1.5 or symptoms of hepatitis worsen (nausea, vomiting, abdominal pain), in which case go to Strategy 3.
2. Stop Pyrazinamide (Z) alone. Observe, measuring transaminases, bilirubin, and INR every 3 days. If transaminases do not fall to < 5x ULN by day 5, or total bilirubin rises >2.0mg/dl (>34 µmol/L), or INR >1.5 or symptoms of hepatitis worsen at any time (nausea, vomiting, abdominal pain), go to Strategy 3.
3. Current standard of care (the current USA CDC guidelines): stop rifampicin (R), isoniazid (H) and Z immediately and add levofloxacin and an aminoglycoside to ethambutol. Restart R (at full dose) once transaminases are <2X ULN and no hepatitis symptoms. If no increase in transaminases after 7 days add isoniazid (at full dose) and stop levofloxacin and aminoglycoside. If transaminases remain normal on full dose R and H, Z was the likely cause and it should not be re-started and treatment duration should be extended to ≥12 months. If transaminases rise ≥ 5x ULN, or ≥3x ULN with symptoms, at any time after re-introduction of R and/or H the physician should stop R and/or H (depending on which was associated with the transaminase rise). If neither R or H can be used, treat with levofloxacin, an aminoglycoside and ethambutol. If R can be used, but not H, treat with R, levofloxacin and ethambutol. If H can be used, but not R, treat with H, levofloxacin and ethambutol.

The primary endpoint is the proportion of time in the 60 days following randomisation during which neither rifampicin nor isoniazid are given (or the subject is dead). For example, if RH is interrupted for 18 days and the participant dies 48 days after randomization, the endpoint will be 50% [(18+(60-48))/60]. Rifampicin and isoniazid are considered critical drugs in early TBM treatment; inability to use these agents (either through bacterial resistance or patient intolerance) is associated with poor outcome. The vast majority of interruptions are expected to be shorter than one month for strategy 3 (standard of care) but as management strategies 1 and 2 delay the time point of the interruption, a longer cut-off of 60 days was chosen.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older)
* HIV-infected
* Clinical diagnosis of TBM (≥5 days of meningitis symptoms, and CSF abnormalities) and anti-tuberculosis chemotherapy either planned or started by the attending physician

Note: Published diagnostic criteria will be applied to all enrolled participants at the end of the study when all mycobacterial culture results are available. The criteria will sub-divide all cases into definite, probable and possible TBM, and those with an alternative diagnosis.

Exclusion Criteria:

* An additional brain infection (other than TBM) confirmed or suspected: positive CSF Gram or India Ink stain; positive blood or CSF Cryptococcal antigen test; cerebral toxoplasmosis suspected and attending physician wants to give anti-toxoplasmosis treatment with anti-tuberculosis treatment
* More than 6 consecutive days of two or more drugs active against M. tuberculosis immediately before screening
* More than 3 consecutive days of any type of orally or intravenously administered corticosteroid immediately before randomisation
* Dexamethasone considered mandatory for any reason by the attending physician
* Dexamethasone considered to be contraindicated for any reason by the attending physician
* Previously been randomised into the trial for a prior episode of TBM
* Lack of consent from the participant or family member (if the participant is incapacitated by the disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Overall survival until 12 months after randomisation | 12 months from randomisation
  The primary endpoint is overall survival, i.e. the time from randomization to death, during a follow-up period of 12 months. Survivors known to be alive at 12 months will be censored at that time-point and subjects who withdrew or were lost to follow-up before 12 months will be censored at the date they were last known to be alive.

SECONDARY OUTCOMES:
Neurological disability at 12 months (modified Rankin score) | at 12 months
  Neurological disability will be assessed by the modified Rankin score (see below) on months 3, 6, 9, 12, 18 and 24 from randomisation. The main endpoint is the 12 month assessment and subjects who died before 12 months will be treated as having a score of 6 ('Dead').
  The Modified Rankin Scale Score Description 0 No symptoms
  1. Minor symptoms not interfering with lifestyle
  2. Symptoms that lead to some restriction in lifestyle, but do not interfere with the patients ability to look after themselves
  3. Symptoms that restrict lifestyle and prevent totally independent living
  4. Symptoms that clearly prevent independent living, although the patient does not need constant care and attention.
  5. Totally dependent, requiring constant help day and night.
  6. Death
Time to new neurological event (defined as a fall in GCS of ≥2 points for ≥48 hours, new focal neurological sign, or new onset of seizures) or death by 12 months | by 12 months
  A neurological event is defined as a fall in Glasgow coma score by ≥2 points for ≥2 days from the highest previously recorded Glasgow coma score (including baseline) or the onset of any of the following clinical adverse events: cerebellar symptoms, focal neurological signs, or onset of seizures.
Rate of neurological IRIS events up to 6 months from randomisation | 6 months from randomisation
  The rate is defined as the number of IRIS events divided by the observed person-time of follow-up in each treatment group.
Time to new AIDS-defining illness or death by 12 months | by 12 months
  AIDS-defining illnesses will be defined as per the WHO classification.
Serious adverse events by 12 months | by 12 months
  Comparison of the frequency of serious adverse events between treatment groups will form an important part of the study analysis.
HIV-associated malignancy by 12 months | by 12 months
  The three major HIV-associated malignancies are Kaposi sarcoma, high grade B-cell non-Hodgkin lymphoma and invasive cervical cancer.
Overall survival | by 24 months
  The main analysis of this trial will be performed at the time point where all randomized subjects have completed 12 months of follow-up. However, all participants will continue to be followed up for 24 months and overall survival will be reported once 24 month follow-up has been completed for all participants.
Neurological disability | by 24 months
  The main analysis of this trial will be performed at the time point where all randomized subjects have completed 12 months of follow-up. However, all participants will continue to be followed up for 24 months and neurological disability will be reported once 24 month follow-up has been completed for all participants.
Time to new AIDS defining event or death | by 24 months
  The main analysis of this trial will be performed at the time point where all randomized subjects have completed 12 months of follow-up. However, all participants will continue to be followed up for 24 months and this outcome will be reported once 24 month follow-up has been completed for all participants.
Rate of HIV-related malignancy | by 24 months
  The main analysis of this trial will be performed at the time point where all randomized subjects have completed 12 months of follow-up. However, all participants will continue to be followed up for 24 months and this outcome will be reported once 24 month follow-up has been completed for all participants.
Recurrence of TBM within 24 months of follow-up | 24 months
  This outcome will be reported once 24 month follow-up has been completed for all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Thwaites, MD, Principal Investigator — University of Oxford, UK
Locations (6):
- Indonesia (3):
  - Cipto Mangunkusumo Hospital, Jakarta
  - Eijkman-Oxford Clinical Research Unit, Jakarta
  - RSUP Persahabatan Hospital, Jakarta
- Vietnam (3):
  - Hospital for Tropical Diseases, Ho Chi Minh City
  - Oxford University Clinical Research Unit, Ho Chi Minh City
  - Pham Ngoc Thach Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
The Oxford University Clinical Research Unit recognizes the ethical obligation to ensure that optimal use is made of the data and specimens that the investigators collect for our research and the value of sharing individual level data. The investigators aim to ensure that data generated from all our research are collected, curated, managed and shared in a way that maximizes their benefit. When sharing data the investigators have an obligation to ensure that the interests of research participants, researchers and other stakeholders are appropriately protected. The Oxford University Clinical Research Unit data sharing policy and the data request form outline the default procedures for data sharing.

REFERENCES:
- [Background] Thwaites GE, van Toorn R, Schoeman J. Tuberculous meningitis: more questions, still too few answers. Lancet Neurol. 2013 Oct;12(10):999-1010. doi: 10.1016/S1474-4422(13)70168-6. Epub 2013 Aug 23. PMID 23972913
- [Background] Kalita J, Misra UK. Outcome of tuberculous meningitis at 6 and 12 months: a multiple regression analysis. Int J Tuberc Lung Dis. 1999 Mar;3(3):261-5. PMID 10094329
- [Background] Thwaites GE, Duc Bang N, Huy Dung N, Thi Quy H, Thi Tuong Oanh D, Thi Cam Thoa N, Quang Hien N, Tri Thuc N, Ngoc Hai N, Thi Ngoc Lan N, Ngoc Lan N, Hong Duc N, Ngoc Tuan V, Huu Hiep C, Thi Hong Chau T, Phuong Mai P, Thi Dung N, Stepniewska K, Simmons CP, White NJ, Tinh Hien T, Farrar JJ. The influence of HIV infection on clinical presentation, response to treatment, and outcome in adults with Tuberculous meningitis. J Infect Dis. 2005 Dec 15;192(12):2134-41. doi: 10.1086/498220. Epub 2005 Nov 15. PMID 16288379
- [Background] Fallon RJ, Kennedy DH. Rapid diagnosis of tuberculous meningitis. J Infect. 1993 Mar;26(2):226. doi: 10.1016/0163-4453(93)93247-2. No abstract available. PMID 8473775
- [Background] STEWART SM. The bacteriological diagnosis of tuberculous meningitis. J Clin Pathol. 1953 Aug;6(3):241-2. doi: 10.1136/jcp.6.3.241. No abstract available. PMID 13084774
- [Background] Thwaites GE, Chau TT, Farrar JJ. Improving the bacteriological diagnosis of tuberculous meningitis. J Clin Microbiol. 2004 Jan;42(1):378-9. doi: 10.1128/JCM.42.1.378-379.2004. PMID 14715783
- [Background] Nhu NT, Heemskerk D, Thu do DA, Chau TT, Mai NT, Nghia HD, Loc PP, Ha DT, Merson L, Thinh TT, Day J, Chau Nv, Wolbers M, Farrar J, Caws M. Evaluation of GeneXpert MTB/RIF for diagnosis of tuberculous meningitis. J Clin Microbiol. 2014 Jan;52(1):226-33. doi: 10.1128/JCM.01834-13. Epub 2013 Nov 6. PMID 24197880
- [Background] Patel VB, Connolly C, Singh R, Lenders L, Matinyenya B, Theron G, Ndung'u T, Dheda K. Comparison of amplicor and GeneXpert MTB/RIF tests for diagnosis of tuberculous meningitis. J Clin Microbiol. 2014 Oct;52(10):3777-80. doi: 10.1128/JCM.01235-14. Epub 2014 Jul 23. PMID 25056328
- [Background] Marais S, Pepper DJ, Schutz C, Wilkinson RJ, Meintjes G. Presentation and outcome of tuberculous meningitis in a high HIV prevalence setting. PLoS One. 2011;6(5):e20077. doi: 10.1371/journal.pone.0020077. Epub 2011 May 19. PMID 21625509
- [Background] Marais S, Pepper DJ, Marais BJ, Torok ME. HIV-associated tuberculous meningitis--diagnostic and therapeutic challenges. Tuberculosis (Edinb). 2010 Nov;90(6):367-74. doi: 10.1016/j.tube.2010.08.006. Epub 2010 Sep 28. PMID 20880749
- [Background] Thwaites G, Fisher M, Hemingway C, Scott G, Solomon T, Innes J; British Infection Society. British Infection Society guidelines for the diagnosis and treatment of tuberculosis of the central nervous system in adults and children. J Infect. 2009 Sep;59(3):167-87. doi: 10.1016/j.jinf.2009.06.011. Epub 2009 Jul 4. PMID 19643501
- [Background] Masur H, Brooks JT, Benson CA, Holmes KK, Pau AK, Kaplan JE; National Institutes of Health; Centers for Disease Control and Prevention; HIV Medicine Association of the Infectious Diseases Society of America. Prevention and treatment of opportunistic infections in HIV-infected adults and adolescents: Updated Guidelines from the Centers for Disease Control and Prevention, National Institutes of Health, and HIV Medicine Association of the Infectious Diseases Society of America. Clin Infect Dis. 2014 May;58(9):1308-11. doi: 10.1093/cid/ciu094. Epub 2014 Feb 27. PMID 24585567
- [Background] Thwaites GE. Advances in the diagnosis and treatment of tuberculous meningitis. Curr Opin Neurol. 2013 Jun;26(3):295-300. doi: 10.1097/WCO.0b013e3283602814. PMID 23493162
- [Background] Ellard GA, Humphries MJ, Allen BW. Cerebrospinal fluid drug concentrations and the treatment of tuberculous meningitis. Am Rev Respir Dis. 1993 Sep;148(3):650-5. doi: 10.1164/ajrccm/148.3.650. PMID 8368635
- [Background] Ruslami R, Ganiem AR, Dian S, Apriani L, Achmad TH, van der Ven AJ, Borm G, Aarnoutse RE, van Crevel R. Intensified regimen containing rifampicin and moxifloxacin for tuberculous meningitis: an open-label, randomised controlled phase 2 trial. Lancet Infect Dis. 2013 Jan;13(1):27-35. doi: 10.1016/S1473-3099(12)70264-5. Epub 2012 Oct 25. PMID 23103177
- [Background] Heemskerk AD, Bang ND, Mai NT, Chau TT, Phu NH, Loc PP, Chau NV, Hien TT, Dung NH, Lan NT, Lan NH, Lan NN, Phong le T, Vien NN, Hien NQ, Yen NT, Ha DT, Day JN, Caws M, Merson L, Thinh TT, Wolbers M, Thwaites GE, Farrar JJ. Intensified Antituberculosis Therapy in Adults with Tuberculous Meningitis. N Engl J Med. 2016 Jan 14;374(2):124-34. doi: 10.1056/NEJMoa1507062. PMID 26760084
- [Background] Tho DQ, Torok ME, Yen NT, Bang ND, Lan NT, Kiet VS, van Vinh Chau N, Dung NH, Day J, Farrar J, Wolbers M, Caws M. Influence of antituberculosis drug resistance and Mycobacterium tuberculosis lineage on outcome in HIV-associated tuberculous meningitis. Antimicrob Agents Chemother. 2012 Jun;56(6):3074-9. doi: 10.1128/AAC.00319-12. Epub 2012 Apr 2. PMID 22470117
- [Background] Thwaites GE, Lan NT, Dung NH, Quy HT, Oanh DT, Thoa NT, Hien NQ, Thuc NT, Hai NN, Bang ND, Lan NN, Duc NH, Tuan VN, Hiep CH, Chau TT, Mai PP, Dung NT, Stepniewska K, White NJ, Hien TT, Farrar JJ. Effect of antituberculosis drug resistance on response to treatment and outcome in adults with tuberculous meningitis. J Infect Dis. 2005 Jul 1;192(1):79-88. doi: 10.1086/430616. Epub 2005 May 20. PMID 15942897
- [Background] Seddon JA, Visser DH, Bartens M, Jordaan AM, Victor TC, van Furth AM, Schoeman JF, Schaaf HS. Impact of drug resistance on clinical outcome in children with tuberculous meningitis. Pediatr Infect Dis J. 2012 Jul;31(7):711-6. doi: 10.1097/INF.0b013e318253acf8. PMID 22411053
- [Background] Torok ME, Farrar JJ. When to start antiretroviral therapy in HIV-associated tuberculosis. N Engl J Med. 2011 Oct 20;365(16):1538-40. doi: 10.1056/NEJMe1109546. No abstract available. PMID 22010921
- [Background] Abdool Karim SS, Naidoo K, Grobler A, Padayatchi N, Baxter C, Gray AL, Gengiah T, Gengiah S, Naidoo A, Jithoo N, Nair G, El-Sadr WM, Friedland G, Abdool Karim Q. Integration of antiretroviral therapy with tuberculosis treatment. N Engl J Med. 2011 Oct 20;365(16):1492-501. doi: 10.1056/NEJMoa1014181. PMID 22010915
- [Background] Havlir DV, Kendall MA, Ive P, Kumwenda J, Swindells S, Qasba SS, Luetkemeyer AF, Hogg E, Rooney JF, Wu X, Hosseinipour MC, Lalloo U, Veloso VG, Some FF, Kumarasamy N, Padayatchi N, Santos BR, Reid S, Hakim J, Mohapi L, Mugyenyi P, Sanchez J, Lama JR, Pape JW, Sanchez A, Asmelash A, Moko E, Sawe F, Andersen J, Sanne I; AIDS Clinical Trials Group Study A5221. Timing of antiretroviral therapy for HIV-1 infection and tuberculosis. N Engl J Med. 2011 Oct 20;365(16):1482-91. doi: 10.1056/NEJMoa1013607. PMID 22010914
- [Background] Blanc FX, Sok T, Laureillard D, Borand L, Rekacewicz C, Nerrienet E, Madec Y, Marcy O, Chan S, Prak N, Kim C, Lak KK, Hak C, Dim B, Sin CI, Sun S, Guillard B, Sar B, Vong S, Fernandez M, Fox L, Delfraissy JF, Goldfeld AE; CAMELIA (ANRS 1295-CIPRA KH001) Study Team. Earlier versus later start of antiretroviral therapy in HIV-infected adults with tuberculosis. N Engl J Med. 2011 Oct 20;365(16):1471-81. doi: 10.1056/NEJMoa1013911. PMID 22010913
- [Background] Torok ME, Yen NT, Chau TT, Mai NT, Phu NH, Mai PP, Dung NT, Chau NV, Bang ND, Tien NA, Minh NH, Hien NQ, Thai PV, Dong DT, Anh DT, Thoa NT, Hai NN, Lan NN, Lan NT, Quy HT, Dung NH, Hien TT, Chinh NT, Simmons CP, de Jong M, Wolbers M, Farrar JJ. Timing of initiation of antiretroviral therapy in human immunodeficiency virus (HIV)--associated tuberculous meningitis. Clin Infect Dis. 2011 Jun;52(11):1374-83. doi: 10.1093/cid/cir230. PMID 21596680
- [Background] Dass R, Nagaraj R, Murlidharan J, Singhi S. Hyponatraemia and hypovolemic shock with tuberculous meningitis. Indian J Pediatr. 2003 Dec;70(12):995-7. doi: 10.1007/BF02723828. PMID 14719791
- [Background] Figaji AA, Fieggen AG. The neurosurgical and acute care management of tuberculous meningitis: evidence and current practice. Tuberculosis (Edinb). 2010 Nov;90(6):393-400. doi: 10.1016/j.tube.2010.09.005. Epub 2010 Oct 20. PMID 20970381
- [Background] Celik U, Celik T, Tolunay O, Baspinar H, Komur M, Levent F. Cerebral salt wasting in tuberculous meningitis: Two cases and review of the literature. Case Report. Neuro Endocrinol Lett. 2015;36(4):306-10. PMID 26454484
- [Background] Pepper DJ, Marais S, Maartens G, Rebe K, Morroni C, Rangaka MX, Oni T, Wilkinson RJ, Meintjes G. Neurologic manifestations of paradoxical tuberculosis-associated immune reconstitution inflammatory syndrome: a case series. Clin Infect Dis. 2009 Jun 1;48(11):e96-107. doi: 10.1086/598988. PMID 19405867
- [Background] Marais S, Wilkinson KA, Lesosky M, Coussens AK, Deffur A, Pepper DJ, Schutz C, Ismail Z, Meintjes G, Wilkinson RJ. Neutrophil-associated central nervous system inflammation in tuberculous meningitis immune reconstitution inflammatory syndrome. Clin Infect Dis. 2014 Dec 1;59(11):1638-47. doi: 10.1093/cid/ciu641. Epub 2014 Aug 8. PMID 25107295
- [Background] Marais S, Meintjes G, Pepper DJ, Dodd LE, Schutz C, Ismail Z, Wilkinson KA, Wilkinson RJ. Frequency, severity, and prediction of tuberculous meningitis immune reconstitution inflammatory syndrome. Clin Infect Dis. 2013 Feb;56(3):450-60. doi: 10.1093/cid/cis899. Epub 2012 Oct 24. PMID 23097584
- [Background] Meintjes G, Wilkinson RJ, Morroni C, Pepper DJ, Rebe K, Rangaka MX, Oni T, Maartens G. Randomized placebo-controlled trial of prednisone for paradoxical tuberculosis-associated immune reconstitution inflammatory syndrome. AIDS. 2010 Sep 24;24(15):2381-90. doi: 10.1097/QAD.0b013e32833dfc68. PMID 20808204
- [Background] Schoeman J, Donald P, van Zyl L, Keet M, Wait J. Tuberculous hydrocephalus: comparison of different treatments with regard to ICP, ventricular size and clinical outcome. Dev Med Child Neurol. 1991 May;33(5):396-405. doi: 10.1111/j.1469-8749.1991.tb14899.x. PMID 2065826
- [Background] Chugh A, Husain M, Gupta RK, Ojha BK, Chandra A, Rastogi M. Surgical outcome of tuberculous meningitis hydrocephalus treated by endoscopic third ventriculostomy: prognostic factors and postoperative neuroimaging for functional assessment of ventriculostomy. J Neurosurg Pediatr. 2009 May;3(5):371-7. doi: 10.3171/2009.1.PEDS0947. PMID 19409015
- [Background] Thwaites GE, Macmullen-Price J, Tran TH, Pham PM, Nguyen TD, Simmons CP, White NJ, Tran TH, Summers D, Farrar JJ. Serial MRI to determine the effect of dexamethasone on the cerebral pathology of tuberculous meningitis: an observational study. Lancet Neurol. 2007 Mar;6(3):230-6. doi: 10.1016/S1474-4422(07)70034-0. PMID 17303529
- [Background] Sheu JJ, Hsu CY, Yuan RY, Yang CC. Clinical characteristics and treatment delay of cerebral infarction in tuberculous meningitis. Intern Med J. 2012 Mar;42(3):294-300. doi: 10.1111/j.1445-5994.2010.02256.x. Epub 2010 May 11. PMID 20492009
- [Background] Shukla R, Abbas A, Kumar P, Gupta RK, Jha S, Prasad KN. Evaluation of cerebral infarction in tuberculous meningitis by diffusion weighted imaging. J Infect. 2008 Oct;57(4):298-306. doi: 10.1016/j.jinf.2008.07.012. Epub 2008 Aug 28. PMID 18760486
- [Background] Springer P, Swanevelder S, van Toorn R, van Rensburg AJ, Schoeman J. Cerebral infarction and neurodevelopmental outcome in childhood tuberculous meningitis. Eur J Paediatr Neurol. 2009 Jul;13(4):343-9. doi: 10.1016/j.ejpn.2008.07.004. Epub 2008 Aug 30. PMID 18757219
- [Background] Koh SB, Kim BJ, Park MH, Yu SW, Park KW, Lee DH. Clinical and laboratory characteristics of cerebral infarction in tuberculous meningitis: a comparative study. J Clin Neurosci. 2007 Nov;14(11):1073-7. doi: 10.1016/j.jocn.2006.07.014. PMID 17954374
- [Background] Schoeman JF, Janse van Rensburg A, Laubscher JA, Springer P. The role of aspirin in childhood tuberculous meningitis. J Child Neurol. 2011 Aug;26(8):956-62. doi: 10.1177/0883073811398132. Epub 2011 May 31. PMID 21628697
- [Background] Misra UK, Kalita J, Nair PP. Role of aspirin in tuberculous meningitis: a randomized open label placebo controlled trial. J Neurol Sci. 2010 Jun 15;293(1-2):12-7. doi: 10.1016/j.jns.2010.03.025. Epub 2010 Apr 24. PMID 20421121
- [Background] Thwaites GE, Nguyen DB, Nguyen HD, Hoang TQ, Do TT, Nguyen TC, Nguyen QH, Nguyen TT, Nguyen NH, Nguyen TN, Nguyen NL, Nguyen HD, Vu NT, Cao HH, Tran TH, Pham PM, Nguyen TD, Stepniewska K, White NJ, Tran TH, Farrar JJ. Dexamethasone for the treatment of tuberculous meningitis in adolescents and adults. N Engl J Med. 2004 Oct 21;351(17):1741-51. doi: 10.1056/NEJMoa040573. PMID 15496623
- [Background] Ramappa V, Aithal GP. Hepatotoxicity Related to Anti-tuberculosis Drugs: Mechanisms and Management. J Clin Exp Hepatol. 2013 Mar;3(1):37-49. doi: 10.1016/j.jceh.2012.12.001. Epub 2012 Dec 20. PMID 25755470
- [Background] Prasad K, Singh MB. Corticosteroids for managing tuberculous meningitis. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD002244. doi: 10.1002/14651858.CD002244.pub3. PMID 18254003
- [Background] Simmons CP, Thwaites GE, Quyen NT, Chau TT, Mai PP, Dung NT, Stepniewska K, White NJ, Hien TT, Farrar J. The clinical benefit of adjunctive dexamethasone in tuberculous meningitis is not associated with measurable attenuation of peripheral or local immune responses. J Immunol. 2005 Jul 1;175(1):579-90. doi: 10.4049/jimmunol.175.1.579. PMID 15972695
- [Background] Tobin DM, Roca FJ, Oh SF, McFarland R, Vickery TW, Ray JP, Ko DC, Zou Y, Bang ND, Chau TT, Vary JC, Hawn TR, Dunstan SJ, Farrar JJ, Thwaites GE, King MC, Serhan CN, Ramakrishnan L. Host genotype-specific therapies can optimize the inflammatory response to mycobacterial infections. Cell. 2012 Feb 3;148(3):434-46. doi: 10.1016/j.cell.2011.12.023. PMID 22304914
- [Background] Tobin DM, Vary JC Jr, Ray JP, Walsh GS, Dunstan SJ, Bang ND, Hagge DA, Khadge S, King MC, Hawn TR, Moens CB, Ramakrishnan L. The lta4h locus modulates susceptibility to mycobacterial infection in zebrafish and humans. Cell. 2010 Mar 5;140(5):717-30. doi: 10.1016/j.cell.2010.02.013. PMID 20211140
- [Background] Prasad K, Singh MB, Ryan H. Corticosteroids for managing tuberculous meningitis. Cochrane Database Syst Rev. 2016 Apr 28;4(4):CD002244. doi: 10.1002/14651858.CD002244.pub4. PMID 27121755
- [Background] Elliott AM, Luzze H, Quigley MA, Nakiyingi JS, Kyaligonza S, Namujju PB, Ducar C, Ellner JJ, Whitworth JA, Mugerwa R, Johnson JL, Okwera A. A randomized, double-blind, placebo-controlled trial of the use of prednisolone as an adjunct to treatment in HIV-1-associated pleural tuberculosis. J Infect Dis. 2004 Sep 1;190(5):869-78. doi: 10.1086/422257. Epub 2004 Jul 29. PMID 15295690
- [Background] Mayosi BM, Ntsekhe M, Bosch J, Pandie S, Jung H, Gumedze F, Pogue J, Thabane L, Smieja M, Francis V, Joldersma L, Thomas KM, Thomas B, Awotedu AA, Magula NP, Naidoo DP, Damasceno A, Chitsa Banda A, Brown B, Manga P, Kirenga B, Mondo C, Mntla P, Tsitsi JM, Peters F, Essop MR, Russell JB, Hakim J, Matenga J, Barasa AF, Sani MU, Olunuga T, Ogah O, Ansa V, Aje A, Danbauchi S, Ojji D, Yusuf S; IMPI Trial Investigators. Prednisolone and Mycobacterium indicus pranii in tuberculous pericarditis. N Engl J Med. 2014 Sep 18;371(12):1121-30. doi: 10.1056/NEJMoa1407380. Epub 2014 Sep 1. PMID 25178809
- [Background] Beardsley J, Wolbers M, Kibengo FM, Ggayi AB, Kamali A, Cuc NT, Binh TQ, Chau NV, Farrar J, Merson L, Phuong L, Thwaites G, Van Kinh N, Thuy PT, Chierakul W, Siriboon S, Thiansukhon E, Onsanit S, Supphamongkholchaikul W, Chan AK, Heyderman R, Mwinjiwa E, van Oosterhout JJ, Imran D, Basri H, Mayxay M, Dance D, Phimmasone P, Rattanavong S, Lalloo DG, Day JN; CryptoDex Investigators. Adjunctive Dexamethasone in HIV-Associated Cryptococcal Meningitis. N Engl J Med. 2016 Feb 11;374(6):542-54. doi: 10.1056/NEJMoa1509024. PMID 26863355
- [Background] Thwaites GE, Bhavnani SM, Chau TT, Hammel JP, Torok ME, Van Wart SA, Mai PP, Reynolds DK, Caws M, Dung NT, Hien TT, Kulawy R, Farrar J, Ambrose PG. Randomized pharmacokinetic and pharmacodynamic comparison of fluoroquinolones for tuberculous meningitis. Antimicrob Agents Chemother. 2011 Jul;55(7):3244-53. doi: 10.1128/AAC.00064-11. Epub 2011 Apr 18. PMID 21502621
- [Background] Meintjes G, Lawn SD, Scano F, Maartens G, French MA, Worodria W, Elliott JH, Murdoch D, Wilkinson RJ, Seyler C, John L, van der Loeff MS, Reiss P, Lynen L, Janoff EN, Gilks C, Colebunders R; International Network for the Study of HIV-associated IRIS. Tuberculosis-associated immune reconstitution inflammatory syndrome: case definitions for use in resource-limited settings. Lancet Infect Dis. 2008 Aug;8(8):516-23. doi: 10.1016/S1473-3099(08)70184-1. PMID 18652998
- [Background] Lokhnygina Y, Helterbrand JD. Cox regression methods for two-stage randomization designs. Biometrics. 2007 Jun;63(2):422-8. doi: 10.1111/j.1541-0420.2007.00707.x. Epub 2007 Apr 9. PMID 17425633
- [Background] Saukkonen JJ, Cohn DL, Jasmer RM, Schenker S, Jereb JA, Nolan CM, Peloquin CA, Gordin FM, Nunes D, Strader DB, Bernardo J, Venkataramanan R, Sterling TR; ATS (American Thoracic Society) Hepatotoxicity of Antituberculosis Therapy Subcommittee. An official ATS statement: hepatotoxicity of antituberculosis therapy. Am J Respir Crit Care Med. 2006 Oct 15;174(8):935-52. doi: 10.1164/rccm.200510-1666ST. PMID 17021358
- [Background] Devarbhavi H, Singh R, Patil M, Sheth K, Adarsh CK, Balaraju G. Outcome and determinants of mortality in 269 patients with combination anti-tuberculosis drug-induced liver injury. J Gastroenterol Hepatol. 2013 Jan;28(1):161-7. doi: 10.1111/j.1440-1746.2012.07279.x. PMID 23020522
- [Background] Pukenyte E, Lescure FX, Rey D, Rabaud C, Hoen B, Chavanet P, Laiskonis AP, Schmit JL, May T, Mouton Y, Yazdanpanah Y. Incidence of and risk factors for severe liver toxicity in HIV-infected patients on anti-tuberculosis treatment. Int J Tuberc Lung Dis. 2007 Jan;11(1):78-84. PMID 17217134
- [Background] Tahaoglu K, Atac G, Sevim T, Tarun T, Yazicioglu O, Horzum G, Gemci I, Ongel A, Kapakli N, Aksoy E. The management of anti-tuberculosis drug-induced hepatotoxicity. Int J Tuberc Lung Dis. 2001 Jan;5(1):65-9. PMID 11263519
- [Background] Sharma SK, Singla R, Sarda P, Mohan A, Makharia G, Jayaswal A, Sreenivas V, Singh S. Safety of 3 different reintroduction regimens of antituberculosis drugs after development of antituberculosis treatment-induced hepatotoxicity. Clin Infect Dis. 2010 Mar 15;50(6):833-9. doi: 10.1086/650576. PMID 20156055
- [Background] Lenaerts A, Barry CE 3rd, Dartois V. Heterogeneity in tuberculosis pathology, microenvironments and therapeutic responses. Immunol Rev. 2015 Mar;264(1):288-307. doi: 10.1111/imr.12252. PMID 25703567
- [Background] Roca FJ, Ramakrishnan L. TNF dually mediates resistance and susceptibility to mycobacteria via mitochondrial reactive oxygen species. Cell. 2013 Apr 25;153(3):521-34. doi: 10.1016/j.cell.2013.03.022. Epub 2013 Apr 11. PMID 23582643
- [Background] Naranbhai V, Moodley D, Chipato T, Stranix-Chibanda L, Nakabaiito C, Kamateeka M, Musoke P, Manji K, George K, Emel LM, Richardson P, Andrew P, Fowler M, Fletcher H, McShane H, Coovadia HM, Hill AV; HPTN 046 Protocol Team. The association between the ratio of monocytes: lymphocytes and risk of tuberculosis among HIV-infected postpartum women. J Acquir Immune Defic Syndr. 2014 Dec 15;67(5):573-5. doi: 10.1097/QAI.0000000000000353. PMID 25247435
- [Background] Naranbhai V, Kim S, Fletcher H, Cotton MF, Violari A, Mitchell C, Nachman S, McSherry G, McShane H, Hill AV, Madhi SA. The association between the ratio of monocytes:lymphocytes at age 3 months and risk of tuberculosis (TB) in the first two years of life. BMC Med. 2014 Jul 17;12:120. doi: 10.1186/s12916-014-0120-7. PMID 25034889
- [Background] Naranbhai V, Hill AV, Abdool Karim SS, Naidoo K, Abdool Karim Q, Warimwe GM, McShane H, Fletcher H. Ratio of monocytes to lymphocytes in peripheral blood identifies adults at risk of incident tuberculosis among HIV-infected adults initiating antiretroviral therapy. J Infect Dis. 2014 Feb 15;209(4):500-9. doi: 10.1093/infdis/jit494. Epub 2013 Sep 16. PMID 24041796
- [Background] Sharma SK, Balamurugan A, Saha PK, Pandey RM, Mehra NK. Evaluation of clinical and immunogenetic risk factors for the development of hepatotoxicity during antituberculosis treatment. Am J Respir Crit Care Med. 2002 Oct 1;166(7):916-9. doi: 10.1164/rccm.2108091. PMID 12359646
- [Background] Hutchings S, Bisset L, Cantillon L, Keating-Brown P, Jeffreys S, Muzvidziwa C, Richmond E, Rees P. Nurse-delivered focused echocardiography to determine intravascular volume status in a deployed maritime critical care unit. J R Nav Med Serv. 2015;101(2):124-8. PMID 26867411
- [Background] Marik PE. Techniques for assessment of intravascular volume in critically ill patients. J Intensive Care Med. 2009 Sep-Oct;24(5):329-37. doi: 10.1177/0885066609340640. PMID 19648183
- [Background] Komut E, Kozaci N, Sonmez BM, Yilmaz F, Komut S, Yildirim ZN, Beydilli I, Yel C. Bedside sonographic measurement of optic nerve sheath diameter as a predictor of intracranial pressure in ED. Am J Emerg Med. 2016 Jun;34(6):963-7. doi: 10.1016/j.ajem.2016.02.012. Epub 2016 Feb 12. PMID 26944107
- [Background] Aduayi OS, Asaleye CM, Adetiloye VA, Komolafe EO, Aduayi VA. Optic nerve sonography: A noninvasive means of detecting raised intracranial pressure in a resource-limited setting. J Neurosci Rural Pract. 2015 Oct-Dec;6(4):563-7. doi: 10.4103/0976-3147.165347. PMID 26752428
- [Background] Dooley KE, Chaisson RE. Tuberculosis and diabetes mellitus: convergence of two epidemics. Lancet Infect Dis. 2009 Dec;9(12):737-46. doi: 10.1016/S1473-3099(09)70282-8. PMID 19926034
- [Background] Pizzol D, Di Gennaro F, Chhaganlal KD, Fabrizio C, Monno L, Putoto G, Saracino A. Tuberculosis and diabetes: current state and future perspectives. Trop Med Int Health. 2016 Jun;21(6):694-702. doi: 10.1111/tmi.12704. Epub 2016 May 18. PMID 27102229
- [Background] Salgame P, Yap GS, Gause WC. Effect of helminth-induced immunity on infections with microbial pathogens. Nat Immunol. 2013 Nov;14(11):1118-1126. doi: 10.1038/ni.2736. PMID 24145791
- [Background] George PJ, Pavan Kumar N, Jaganathan J, Dolla C, Kumaran P, Nair D, Banurekha VV, Shen K, Nutman TB, Babu S. Modulation of pro- and anti-inflammatory cytokines in active and latent tuberculosis by coexistent Strongyloides stercoralis infection. Tuberculosis (Edinb). 2015 Dec;95(6):822-828. doi: 10.1016/j.tube.2015.09.009. Epub 2015 Oct 8. PMID 26542223
- [Derived] Donovan J, Bang ND, Imran D, Nghia HDT, Burhan E, Huong DTT, Hiep NTT, Ngoc LHB, Thanh DV, Thanh NT, Wardhani ALS, Maharani K, Gasmara CP, Hanh NHH, Oanh PKN, Estiasari R, Thu DDA, Kusumaningrum A, Dung LT, Giang DC, Ha DTM, Lan NH, Chau NVV, Nguyet NTM, Geskus RB, Thuong NTT, Kestelyn E, Hamers RL, Phu NH, Thwaites GE; ACT HIV Investigators. Adjunctive Dexamethasone for Tuberculous Meningitis in HIV-Positive Adults. N Engl J Med. 2023 Oct 12;389(15):1357-1367. doi: 10.1056/NEJMoa2216218. PMID 37819954
- [Derived] Donovan J, Oanh PKN, Dobbs N, Phu NH, Nghia HDT, Summers D, Thuong NTT, Thwaites GE; Vietnam ICU Translational Applications Laboratory (VITAL) Investigators. Optic Nerve Sheath Ultrasound for the Detection and Monitoring of Raised Intracranial Pressure in Tuberculous Meningitis. Clin Infect Dis. 2021 Nov 2;73(9):e3536-e3544. doi: 10.1093/cid/ciaa1823. PMID 33283229